CLINICAL TRIAL: NCT06012097
Title: Impact of Gel Aromatherapy on Pain for Patients With De Quervain Disease : Monocentric Study, Controlled, Randomized, Partially Blinded, in Paralleled Groups
Brief Title: Impact of Gel Aromatherapy on Pain for Patients With De Quervain Disease
Acronym: Helping Hand
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7452
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: De Quervain Disease
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active comparator (Active Comparator): Diclofenac gel Splint of the thumb and wrist
  Interventions: Drug: Diclofenac gel
- Experimental Group (Experimental): Aromatherapy Gel Splint of the thumb and wrist
  Interventions: Drug: Aromatherapy gel

INTERVENTIONS:
Drug: Diclofenac gel — using diclofenac as a comparator
  Arms: active comparator
Drug: Aromatherapy gel — using Aromatherapy gel as an experimetnal treatment
  Arms: Experimental Group

SUMMARY:
De Quervain disease is characterized by an adductor pollicis longus and extensor pollicis brevis tendons inflammation as thys pass beneath the extensor retinaculum at the radial styloid. This pathology is recognized as a musculoskeletal disorder of the upper limb triggering functional deficits resulting to possible modifications in the professional activity, sources of absenteeism, thus constituting an economic cost for society. At the etiological level, this pathology also affects young mothers (it's called "mother's wrist" or mommy thumb"), mobile phone users ("textonite", "Blackberryte") or video game players ("Nintendoite").

Currently, the treatment is mainly conservative by splint and anti-inflammatory gel and/or corticosteroid infiltration. Howewer, these therapies have undesirable effects. The interest of this study is therefore to propose another therapy based on aromatherapy gel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 to 75,
* Patient with unilateral De Quervain's tenosynovitis,
* Patient cared in the Hand Surgery Department, SOS Mains Emergency Department or Rheumatology Department of Strasbourg University Hospitals,
* Patient informed of the results of the prior medical examination,
* Informed consent signed by the patient,
* Patient affiliated to a health insurance social protection scheme or beneficiary,
* For a woman of childbearing potential, negative urine pregnancy test at the inclusion visit and maintenance of effective contraception throughout the study.

Exclusion Criteria:

* Pregnant or breastfeeding patient,
* Patient allergic to a component of the gel with essential oils, Dicloflenac®, NSAIDs, or one of the excipients
* Patient treated with oral non-steroidal anti-inflammatory drugs
* Patient with ongoing treatment with another ointment at the treatment application site (radial edge of the wrist)
* Patient with damaged skin, whatever the lesion: oozing dermatosis, eczema, infected lesion, burn or wound,
* Patient with atopic skin disease,
* Patient with epilepsy or with a history of epilepsy,
* Patient with a history of homolateral De Quervain's tenosynovitis, or having already had corticosteroid infiltrations in the 6 months before his inclusion on the ipsilateral side of the pathology,
* Patient with associated tendinopathies in the elbow or forearm region,
* Impossibility of giving the patient information (patient in an emergency situation, patient with difficulties of understandin, agitation of the patient),
* Patient under legal protection, under guardianship or curatorship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Measure of pain during the WHAT test | Day 0
  Visual analogue pain scale (quotation between 0 and 10) during WHAT Test
Measure of pain during the WHAT test | Day 42
  Visual analogue pain scale (quotation between 0 and 10) during WHAT Test
Measure of pain during the WHAT test | Day 84
  Visual analogue pain scale (quotation between 0 and 10) during WHAT Test

CONTACTS AND LOCATIONS:
Locations (1):
- Service SOS Main, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No